CLINICAL TRIAL: NCT06146465
Title: Mobile Health Applications in Pediatric Patient Management: Clinicians' Perceptions, Expectations and Experiences
Status: Recruiting | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Derşan Onur, Principal Investigator, Dr. Behcet Uz Children's Hospital
Other Study IDs: Pediatric mHealth
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Mobile Health; Pediatrics
Keywords: mobile health; pediatric

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatrics: attending and resident pediatrics physicians involved in pediatric patient management
  Interventions: Other: speciality
- Non-Pediatrics physicians: attending and resident non-pediatrics physicians involved in pediatric patient management
  Interventions: Other: speciality

INTERVENTIONS:
Other: speciality — Not

SUMMARY:
The goal of this observational study is to to determine the perceptions, expectations and experiences of physicians involved in pediatric patient management about mHealth applications. The main questions it aims to answer are:

* Is the use of mHealth applications in pediatric patient management different between pediatricians and other specialties?
* What are the most commonly used mHealth applications in pediatric patient management? Participants will fill out an online survey form.

DETAILED DESCRIPTION:
With the development of mobile devices, applications that have become widely used have also affected the provision of healthcare services. Efficient and fast applications that can be used by healthcare professionals as well as patients have begun to be developed. This has been shaped in different aspects by information and time management, calculations, communication, consultancy, electronic health record, patient management and monitoring, medical education and training, decision support system, reference and search for updated information.

There are many studies on physicians' use of mHealth applications. However, each clinic and each medical branch will have different expectations from mHealth applications. The investigators do not know the applications used by physicians participating in pediatric patient management in our country, their expectations from these applications, and their solutions. The investigators aim to learn the perceptions, expectations and experiences of physicians involved in pediatric patient management in Turkey about mHealth applications, and thus to guide future mHealth applications from the perspective of child health and diseases.

An online survey will be used as a data collection tool in our research. The online survey method was preferred in order to keep the research population and sample wide.

Our survey will consist of four sections and a total of 28 questions. Survey questions were derived by reviewing previous studies and national clinical experience. In the pilot study, 10 clinicians were asked to complete the survey. Feedback was received on the operation, duration, structure and readability of the questions of the survey. To ensure content validity and reliability, our survey was revised after the ethics committee evaluation and feedback given through the pilot application.

The first part was about physicians' basic demographic data and mobile device usage. Clinicians' perceptions regarding mHealth application usage were evaluated in the second section, their experiences were evaluated in the third section, and their expectations were evaluated in the fourth section. Those who did not agree to participate in the survey were asked a multiple-choice question asking why. Multiple choice, ranking, five-point Likert scale, and free text (age, etc.) questions were used in the survey. Additionally, in order to increase the reliability of the survey, some control questions were designed as negative-positive questions.

Our study will be reported in accordance with the CROSS (A Consensus-Based Checklist for Reporting of Survey Studies) guideline.

ELIGIBILITY:
Inclusion Criteria:

* Being a medical doctor involved in the management of pediatric patients (0-18 years old)

Exclusion Criteria:

* Other specialists outside of pediatrics and family medicine.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Our research population consists of approximately 8500 physicians for pediatricians, approximately 25000 physicians for family physicians, and 15000 physicians for general practitioners in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of clinicians' use of mHealth applications | 12/01/2023-01/01/2024
  How often is it used per week?
duration of clinicians' use of mHealth applications | 12/01/2023-01/01/2024
  How long do they use it?

CONTACTS AND LOCATIONS:
Overall Officials: Derşan Onur, Principal Investigator — Dr. Behcet Uz Children's Hospital
Locations (1):
- Dr. Behcet Uz Children's Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El Hadidy TS, Alshafei AE, Mortell AE, Doherty EM. Smartphones in clinical practice: doctors' experience at two Dublin paediatric teaching hospitals. Ir J Med Sci. 2018 Aug;187(3):565-573. doi: 10.1007/s11845-017-1713-x. Epub 2017 Nov 23. PMID 29170970
- [Result] Jahn HK, Jahn IHJ, Behringer W, Lyttle MD, Roland D; Paediatric Emergency Research United Kingdom and Ireland (PERUKI). A survey of mHealth use from a physician perspective in paediatric emergency care in the UK and Ireland. Eur J Pediatr. 2021 Aug;180(8):2409-2418. doi: 10.1007/s00431-021-04023-0. Epub 2021 Mar 25. PMID 33763717
- [Result] Hadjipanayis A, Klonis A, Abdel-Mannan OA, Sutcliffe AG. Smartphone use in Paediatric Practice: a national survey. J Mob Technol Med. 2016;5(1):3-8. doi:10.7309/jmtm.5.1.2